CLINICAL TRIAL: NCT05146674
Title: Impact of Tadalafil 5 mg on Post-micturition Dribble in Young-age Men With no/Mild Lower Urinary Tract Symptoms: a Randomized Controlled Trial
Brief Title: Impact of Tadalafil 5 mg on Post-micturition Dribble in Young-age Men With no/Mild Lower Urinary Tract Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Lecturer of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AS-11-2021
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Post-micturition dribble; Lower urinary tract symptoms; Tadalafil; Quality of life
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil group (Active Comparator): Our prospective, randomized, study will consist of a 1-week baseline period and 12-week double-blind treatment period During the baseline period, patients' characteristics, including medical and sexual history, physical examination results, vital signs, HPMDQ score, IPSS, International Index of Erectile Function (IIEF) score, PMD volume, and uroflowmetry results; and laboratory results, including urine analysis results, will be recorded.
  After the baseline period, patients will be randomly assigned, 1:1, to the treatment or control groups using a computer-generated system. Both study groups will be advised to do bulbar urethral massage in addition to pelvic floor muscle exercise (explained later) during the study period, treatment group will be given tadalafil 5 mg (treatment group) daily or no medication (control group).
  Interventions: Drug: Tadalafil 5mg
- Control group (No Intervention): Our prospective, randomized, study will consist of a 1-week baseline period and 12-week double-blind treatment period During the baseline period, patients' characteristics, including medical and sexual history, physical examination results, vital signs, HPMDQ score, IPSS, International Index of Erectile Function (IIEF) score, PMD volume, and uroflowmetry results; and laboratory results, including urine analysis results, will be recorded.
  After the baseline period, patients will be randomly assigned, 1:1, to the treatment or control groups using a computer-generated system. Both study groups will be advised to do bulbar urethral massage in addition to pelvic floor muscle exercise (explained later) during the study period, treatment group will be given tadalafil 5 mg (treatment group) daily or no medication (control group).

INTERVENTIONS:
Drug: Tadalafil 5mg — Our prospective, randomized, study will consist of a 1-week baseline period and 12-week double-blind treatment period During the baseline period, patients' characteristics, including medical and sexual history, physical examination results, vital signs, HPMDQ score, IPSS, International Index of Erectile Function (IIEF) score, PMD volume, and uroflowmetry results; and laboratory results, including urine analysis results, will be recorded.
  After the baseline period, patients will be randomly assigned, 1:1, to the treatment or control groups using a computer-generated system. Both study groups will be advised to do bulbar urethral massage in addition to pelvic floor muscle exercise (explained later) during the study period, treatment group will be given tadalafil 5 mg (treatment group) daily or no medication (control group).
  Arms: Tadalafil group

SUMMARY:
The primary objective of this prospective, single-centre randomized controlled trial is to assess the efficacy of tadalafil 5 mg on post-micturition dribble (PMD) in young age men (18-50 years) with no/mild lower urinary tract symptoms (LUTS).

DETAILED DESCRIPTION:
Post-micturition dribble (PMD), a post-voiding symptom, is defined as involuntary loss of urine immediately after urination. It is more common in males. Many population/practice-based studies have shown that PMD is one of the most common bothersome urinary symptoms in adult males ranging from 5.5 % to 29 %. (1, 2) In young age men (less than 50 years) with absence of prostate-associated lower urinary tract symptoms (LUTS), PMD is considered the most devastating urinary complaint with worsened physical and mental health-related quality of life (HRQoL). (3) Pathophysiology of PMD is usually attributed to residual urine in the bulbar urethra whatever the cause. Many theories, including weakness or failure of the pelvic floor muscles, incompetency of the external urethral sphincter or bladder neck obstruction, were suggested for this urine residue. (4) However, in patients with PMD with no/mild LUTS, pelvic floor muscle weakness especially the bulbocavernosus and ischiocavernosus muscles is usually the main putative mechanism. (5) Bulbar urethral massage and pelvic floor muscle exercise have been proposed as useful options for patients with PMD (6); yet, pharmacological treatment has not been standardized for those patients.

In this perspective, recent studies have shown that corpus cavernosum structural changes may be related to PMD. (7) It is well known that phosphodiesterase-5 (PDE-5) isoenzymes are highly expressed in the urethra as well as the corpus cavernosum, bladder and prostate. (8) In addition, once-daily 5 mg tadalafil, a PDE-5 inhibitor, has previously been used to treat voiding and storage LUTS. In addition, tadalafil once daily showed reduced PMD symptom severity and PMD volume in men with PMD and other LUTS. (9) Notably, this study included old age men (mean age 62 years) with moderate or severe LUTS.

The aim of the present study was to compare the effects of taking tadalafil 5 mg once daily on PMD in young men (18-50 years) with minimal/mild LUTS.

ELIGIBILITY:
Inclusion Criteria:

* 1- Adult patients (aged 19-50 years) 2- Complaining from PMD with no or mild LUTS (IPSS<8).

Exclusion Criteria:

* 1- Patients with penile or urethral malformations 2- Patients recently received PDE5Is in the last 4 weeks prior to study start. 3- Systemic illness 4- Contraindications to PDE5Is. 5- History of pelvic surgery or irradiation 6- History of bladder or prostate surgery 7- Other acute medical conditions as acute gastroenteritis, osetoarthritis that might influence the patient QoL

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of post-micturition dribble | 12 weeks
  Improvement of PMD is defined as improvement by Hallym Post-Micturation Dribble Questionnaire (HPMDQ) score will decrease by 2 points or more

SECONDARY OUTCOMES:
Post micturition dribble volume | 12 weeks
  Impact of treatment on PMD volume
Erectile function | 12 weeks
  Impact of treatment on erectile function as assessed by international index of erectile function (IIEF)
Lower urinary tract symptoms | 12 weeks
  Impact of treatment on LUTS as assessed by International prostate symptoms score (IPSS)

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, DK, Egypt